## **Study Title: LA-CEAL 4.0: Wearable Sensor Project**

## **NCT Number**

NCT06086028

Statistical Analysis Plan Date: 11/20/2023

**LA-CEAL 4.0:** Wearable Sensor Project Analysis Plan. Analyses for the primary outcome will test the between group differences in the percentage of days participants reported concordance between high levels of stress and engaging in a self-care activity across immediate and delayed information release arms. Secondary outcomes will test between group differences in the average levels of self-reported burnout, depression, anxiety, and resilience; as well as differences in measurements recorded via wearable sensor such as respiratory rate, activity level, sleep efficiency score, heartrate variability and heartrate (measured as beats per minute). Analyses will use both paired and independent samples t-test as appropriate. We will also test for statistically significant between groups differences in baseline characteristics.